CLINICAL TRIAL: NCT00780234
Title: Pioglitazone for Lung Cancer Chemoprevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLIN-005-08S
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer; Endobronchial Dysplasia
Keywords: chemoprevention; lung cancer; pioglitazone
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: pioglitazone (Experimental): Current or former smokers receive 6 months of treatment with pioglitazone
  Interventions: Procedure: fluorescence bronchoscopy; Procedure: quantitative high resolution CT scan; Drug: PIOGLITAZONE VS. PLACEBO 30 mg
- Arm 2: placebo (Placebo Comparator): Current or former smokers receive 6 months of treatment with placebo
  Interventions: Procedure: fluorescence bronchoscopy; Procedure: quantitative high resolution CT scan

INTERVENTIONS:
Procedure: fluorescence bronchoscopy — examination of the central airways with a bronchoscope. Both white light and fluorescent light will be used.
Procedure: quantitative high resolution CT scan — High resolution CT scan of the chest
Drug: PIOGLITAZONE VS. PLACEBO 30 mg — Patients will be randomized to receive either pioglitazone or placebo. Pioglitazone hydrochloride, a thiazolidinedione antidiabetic agent and a potent peroxisome proliferator-
  activated receptor-gamma agonist. It is FDA approved for the treatment of Type II diabetes. It has been previously administered to non-diabetic subjects. The most common side effect of pioglitazone is fluid retention and modest weight gain. There is a potential risk that pioglitazone may cause an elevation in liver enzymes and more serious hepatotoxicity (rare). There is risk of edema and weight gain associated with pioglitazone therapy. 5% experienced peripheral edema in clinical trials. fluid retention may result in new onset heart failure or exacerbation of existing heart failure. Small risk of hypoglycemia, anemia, myalgia, bone fracture, headache, and macular retinal edema exists. There is insufficient information to confirm its safety in Pregnancy/Breastfeeding. Bladder cancer is more serious but rare.
  Arms: Arm 1: pioglitazone

SUMMARY:
This is a chemoprevention trial evaluating the diabetic agent pioglitazone. Non-diabetic subjects at risk for lung cancer (based on smoking history, lung function testing, and atypical cells in a sputum sample) receive either placebo or pioglitazone and have chest computerized tomography (CAT) scans and examinations of their airways with a bronchoscope at the start of the trial and after 6 months on treatment. Compensation will be provided to the subject after completing the trial.

DETAILED DESCRIPTION:
This trial evaluates the oral peroxisome proliferator-activated receptor gamma (PPARgamma) agonist pioglitazone in a double-blind placebo controlled trial. The high risk current and former smokers qualify based on tobacco exposure, airflow limitation on lung function testing, and sputum cytologic atypia. Subjects have a quantitative high resolution thoracic CT scan and a fluorescent bronchoscopy at study entry and after 6 months on drug or placebo. Biologic samples are collected at both time points. The primary outcome is endobronchial histology and determining if pioglitazone can retard progression. Secondary endpoints related to the PPAR gamma signaling pathway will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smoker (at least 10 pack years);
* One or more of the following:
* Mild or worse sputum atypia
* Airflow Limitation (FEV1/FVC<70% predicted)
* Biopsy proven airway dysplasia

Exclusion Criteria:

* myocardial infarction (MI) with ejection fraction < 50%;
* severe/unstable angina;
* history of coronary or peripheral arterial bypass grafting;
* New York Heart Association (NYHA) class III or IV congestive heart failure;
* hypoxemia (less than POX 90 with supplemental oxygen); Diabetes type I or II; severe COPD (GOLD stage III or IV); clinically significant edema requiring diuretic therapy;
* life expectancy < 6 months; history of bladder cancer
* pregnant or breast feeding; inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Keith, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver, CO
Locations (2):
- United States (2):
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Oral iloprost improves endobronchial dysplasia in former smokers — http://www.ncbi.nlm.nih.gov/pubmed/21636546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 243 subjects were consented to provide a pre-screening sputum cytology specimen, and of those, 92 enrolled onto full trial.
Pre-assignment Details: 243 subjects were consented to provide a pre-screening sputum cytology specimen, and of those, 92 enrolled onto full trial.
Groups:
- Arm 1: Pioglitazone: Current or former smokers receive 6 months of treatment with pioglitazone.
  fluorescence bronchoscopy: examination of the central airways with a bronchoscope. Both white light and fluorescent light.
  quantitative high resolution CT scan: High resolution chest CT scan
  PIOGLITAZONE VS. PLACEBO 30 mg: Patients will be randomized to receive either pioglitazone or placebo. Pioglitazone hydrochloride, a thiazolidinedione antidiabetic agent and a potent peroxisome proliferator- activated receptor-gamma agonist.
Period: Overall Study
Arm/Group | Arm 1: Pioglitazone | Arm 2: Placebo
Started | 47 | 45
Completed | 39 | 37
Not Completed | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Pioglitazone: Current or former smokers receive 6 months of treatment with pioglitazone
  fluorescence bronchoscopy: examination of the central airways with a bronchoscope. Both white light and fluorescent light will be used.
  quantitative high resolution CT scan: High resolution CT scan of the chest
  PIOGLITAZONE VS. PLACEBO 30 mg: Patients will be randomized to receive either pioglitazone or placebo. Pioglitazone hydrochloride, a thiazolidinedione antidiabetic agent and a potent peroxisome proliferator-
  activated receptor-gamma agonist. It is FDA approved for the treatment of Type II diabetes. It has been previously administered to non-diabetic subjects. The most common side effect of pioglitazone is fluid retention and modest weight gain. There is a potential risk that pioglitazone may cause an elevation in liver enzymes and more serious hepatotoxicity (rare). There is risk of edema and weight gain associated with pioglitazone therapy. 5% experienced peripheral edema in clinical trials.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pioglitazone | Arm 2: Placebo | Total
Number analyzed (Participants) | 47 | 45 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (9.6) | 62.6 (8.2) | 60.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 39 | 38 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: Hispanic | 4 | 2 | 6
  Ethnicity/Race: Non-Hispanic White | 41 | 36 | 77
  Ethnicity/Race: Non-Hispanic Black | 2 | 6 | 8
  Ethnicity/Race: Non-Hispanic American Indian | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 6-month Histology Score
Description: Biopsies were classified into one of the following 8 World Health Organization defined categories to classify the endobronchial lesion and assign a score according to the following scale: 1 = normal bronchial epithelium; 2 = reserve cell hyperplasia; 3 = squamous metaplasia without atypia; 4 = mild dysplasia; 5 = moderate dysplasia; 6 = severe dysplasia; 7 = carcinoma in situ (CIS); and 8 = invasive carcinoma. 1 represents the best outcome and 8 represents the worst outcome.
Time Frame: 6 months
Population: Although 76 subjects had a 6-month bronchoscopy (39 pioglitazone, 37 placebo), only 64 subjects (34 pioglitazone, 30 placebo) had matched biopsy pairs with non-normal tissue at baseline. Of these 64, 29 were former smokers (15 pioglitazone, 14 placebo), which was the a priori group for the primary analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1: Pioglitazone | Arm 2: Placebo
Number analyzed (Participants) | 15 | 14
Units on a scale | 3.07 (2.02) | 3.71 (2.02)
Statistical Analysis 1: Comparison: Arm 1: Pioglitazone vs Arm 2: Placebo; The hypotheses tested were: H0: α1 = 0 vs H1: α1 ~= 0; Test type: Other; p = 0.53, Regression, Linear; The estimates of treatment effect were adjusted for baseline histology values; Regression model parameter (α1) = -0.40, 95% CI 2-sided [-1.68 to 0.89], Standard Error of Mean 0.63; The hypothesis test was a 2-sided t-test of the effect of group (i.e. the difference between the pioglitazone and placebo groups). The general form of the model is Y = α0 + α1GROUP + α2BASELINE. Y represents the 6-month value of the dependent variable (summary of the histology), GROUP represents a classification variable for the treatment group (1=pioglitazone, 2=placebo), BASELINE represents the value of the outcome measure at baseline, and α0, α1 and α2 represent the parameter estimates from the general linear model. The test of the difference between groups will be the formal test of significance of the α1 parameter

ADVERSE EVENTS:
Time Frame: 4 years, 11 months
Arm/Group | Arm 1: Pioglitazone | Arm 2: Placebo
All-Cause Mortality (participants affected / at risk) | 1/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/47 | 5/45
Other Adverse Events (participants affected / at risk) | 44/47 | 41/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pioglitazone (N=47) | Arm 2: Placebo (N=45)
Alcohol Intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Skin Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Weight Gain (Investigations) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Pioglitazone (N=47) | Arm 2: Placebo (N=45)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 | 28
Hypertension (Cardiac disorders) | 24 | 21
Weight Gain (Investigations) | 20 | 10
Hypocalcemia (Metabolism and nutrition disorders) | 13 | 9
Anemia (Blood and lymphatic system disorders) | 11 | 9
Aspartate Aminotransferase Increased (Investigations) | 11 | 8
Edema Limbs (General disorders) | 6 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 8 | 3
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 6 | 4
GGT Increased (Investigations) | 4 | 7
Alanine Aminotransferase Increased (Investigations) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5
White Blood Cell Decreased (Investigations) | 6 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Sinus Tachycardia (Cardiac disorders) | 5 | 4
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5
Non-Cardiac Chest Pain (General disorders) | 4 | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Fever (General disorders) | 2 | 4
Platelet Count Decreased (Investigations) | 2 | 4
Vomiting (Gastrointestinal disorders) | 3 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Alkaline Phosphatase Increased (Investigations) | 2 | 3
Fatigue (General disorders) | 2 | 3
Dizziness (Nervous system disorders) | 4 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes